CLINICAL TRIAL: NCT02013297
Title: Hypofractionated Stereotactic Radiation Treatments (SBRT) on Children, Teenagers and Young Adults Malignant Tumors
Brief Title: Study of SBRT Efficacy on Intra and Extra -Cranial Tumors or Metastasis in Pediatrics Population (SBRT Pediatrics)
Acronym: SBRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT
Record Dates: First submitted 2013-12-05; First posted 2013-12-17 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Brain Metastasis; Spinal Tumors; Lung Tumors; Ependymoma
Keywords: Pediatrics; SBRT; Brain metastasis; Pulmonary metastasis; Spinal metastasis; Pulmonary primary tumor; Spinal primary tumor; Relapsed ependymoma; Relapsed irradiated tumors; Local control rate; Safety; Overall survival; Progression Free Survival
MeSH Terms: conditions — Brain Neoplasms; Spinal Cord Neoplasms; Lung Neoplasms; Ependymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT treatment (Experimental): According to the site to irradiate and to local constraints, SBRT consist in 1 to 8 fractions of 5 to 18 Gy
  Interventions: Radiation: SBRT treatment

INTERVENTIONS:
Radiation: SBRT treatment — For Brain metastasis the SBRT treatment consists on 3 fractions of 8 Gy or 5 fractions of 7 Gy or 1 fraction of 18 Gy for a single metastasis which is less than 20 mm.
  For primary or secondary pulmonary tumors the SBRT treatment consists on 3 fractions of 15 Gy or 5 fractions of 10 Gy for peripheral lesions and on 5 fractions of 8 Gy for proximal lesions.
  For primary or secondary spinal or para-spinal tumors the SBRT treatment consists on 3 fractions of 9 Gy or 5 fractions of 7 Gy.
  For previously irradiated tumors (same locations) the SBRT treatment consists on 5 to 8 fractions of 5 Gy.
  For relapsed Ependymoma previously irradiated the SBRT treatment will be allocated by surgical stratified randomization and consists on either 3 fractions of 8 Gy or 5 fractions of 5 Gy.

SUMMARY:
The purpose of this study is to evaluate the efficacy of hypofractionated stereotactic radiation treatments (SBRT) on children, teenagers and young adults malignant tumors.

DETAILED DESCRIPTION:
SBRT (Stereotactic Body Radiation Therapy) is a radiotherapy treatment which involves the delivery of a single high dose radiation treatment or a few fractionated radiation treatments (usually up to 5). A high potent biological dose of radiation is delivered to the tumor improving the cure rates for the tumor, in a manner previously not achievable by standard conventional radiation therapy.

For adult patients, the "Haute Authorité de Santé" (HAS) validates some indications for this treatment which are the followings :

* Few primary or secondary brain tumors, which cannot be surgically removed
* Spinal tumors
* Primary bronchopulmonary tumors T1 T2 N0 M0 and pulmonary metastasis with slow growth and controled primary tumor.

For pediatrics patients, no indication is now validated by HAS. Indications validated for adults are rare in pediatrics but not exceptional, and in such cases efficient alternative treatments does not exist.

In consequence, and regarding the good results obtained in adult patients, it seems very important to validate the efficacy of this treatment on pediatrics population

ELIGIBILITY:
INCLUSION CRITERIA:

* 18 months ≤ age ≤ 20 years
* Malignant primary tumor, histologically or cytologically proven
* Systemic disease under control or with slow evolution
* Written indication of SBRT according to local pediatrics meeting and national Radiotherapy (RT) web conference
* Performance Status ≤ 2 according to Eastern Cooperative Oncology Group (ECOG)
* Sites

  * Brain metastasis (≤ 3 on MRI) not suitable for surgery, without hemorrhage, less than 3 cm each, not in the brain stem
  * Primary or secondary spinal/para spinal metastasis (≤ 3), not suitable for surgery or with a non operable macroscopic residue, less than 5 cm
  * Lung metastasis (≤ 3), less than 5 cm, not eligible for surgery, or macroscopic residue not suitable for surgery
  * Previously irradiated relapsing isolated primitive/secondary tumor (intra cranial or extra cranial), with no possible surgery, or macroscopic residue.
* Affiliation to a social security scheme
* Signed Informed consent by patient or parents and patient

IN ADDITION FOR RELAPSING EPENDYMOMA:

* Histologically proven local ependymoma at diagnosis
* Previously irradiated ependymoma
* Exclusive local relapse in previously irradiated site
* Review of operability at time of relapse by a multidisciplinary staff
* Relapse must be confirmed by a neuro-oncology multidisciplinary staff, on MRI evolutivity characteristics
* Time to relapse after previous irradiation ≥ 1 year

NON-INCLUSION CRITERIA :

* Concomitant chemotherapy
* No evaluable target (except for completely resected ependymomas)
* Pregnancy
* Follow-up impossible

IN ADDITION FOR RELAPSING EPENDYMOMAS:

* Metastatic patient at diagnosis and/or at relapse
* Complete remission never obtained

NON-RANDOMIZATION DOSIMETRIC CRITERIA (ONLY FOR EPENDYMOMA)

* Cumulative doses to brain stem ≥ 115 Gy
* Tumor volume at relapse ≥ 30 cm3
* Primary RT dose + Re-irradiation dose more than 112 Gy
* Cumulative dose to the chiasma > 54 Gy
* Cumulative dose to any point of the brain > 115 Gy

Ages: 18 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of SBRT assessed 6 months after treatment | 6 months after inclusion
  The treatment efficacy is assessed by calculation of local control rate of irradiated locations according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria (complete response + partial response + stable disease)

SECONDARY OUTCOMES:
Efficacy of SBRT assessed between 1,5 and 3 months after treatment | Between 1,5 and 3 months after inclusion
  The treatment efficacy is assessed by calculation of local control rate of irradiated locations according to RECIST version 1.1 criteria (complete response + partial response + stable disease) between 1,5 and 3 months after treatment
Progressive Free Survival | From the date of inclusion to the date of progression
  Calculated from the date of inclusion to the date defined as the first documented disease progression, or second cancer appearance, or death from any cause (Up to 5 years since the first inclusion)
Overall Survival | From the date of inclusion to the date of death (Up to 5 years since the first inclusion)
  Calculated from the date of inclusion to the date of death from any cause (Up to 5 years since the first inclusion)
Short time Safety profile of SBRT | From inclusion to 3 months after inclusion
  Toxicities appeared during SBRT treatment and up to 3 months after SBRT. Toxicities will be assessed by the evaluation of intensity and incidence of the Adverse Events (AE) displayed by patients. The intensity of each AE will be classified according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Long term Safety profile of SBRT | after 24 months after inclusion
  Toxicities appeared after 24 months after inclusion. The outcome measure concerns toxicities appeared after the study following period. Toxicities will be assessed by the evaluation of intensity and incidence of the Adverse Events (AE) displayed by patients. The intensity of each AE will be classified according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Efficacy of SBRT assessed 12 months after treatment | 12 months after inclusion
  The treatment efficacy is assessed by calculation of local control rate of irradiated locations according to RECIST version 1.1 criteria (complete response + partial response + stable disease) at 12 months after treatment
Efficacy of SBRT assessed 24 months after treatment | 24 months after inclusion
  The treatment efficacy is assessed by calculation of local control rate of irradiated locations according to RECIST version 1.1 criteria (complete response + partial response + stable disease) at 24 months after treatment
Medium time Safety profile of SBRT | Between 3 months and 24 months after inclusion
  Toxicities appeared between 3 months and 24 months after treatment. Toxicities will be assessed by the evaluation of intensity and incidence of the Adverse Events (AE) displayed by patients. The intensity of each AE will be classified according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

OTHER OUTCOMES:
SBRT treatment and toxicities related costs for 6 months after SBRT | 6 months after inclusion
  The SBRT treatment related costs will be evaluated by a "microcosting" method which take into account, in particular, the irradiation duration seance, the time for the mobilized staff, the kind of equipment required, the duration of related AE hospitalizations.
Cost/Efficacy ratio between 2 modalities of SBRT treatment of ependymoma at 6 months after treatment | 6 months after inclusion
  2 modalities of SBRT are compared in patients with an ependymoma (3 fractions of 8 Gy versus 5 fractions of 5 Gy). It will be calculated the cost/efficacity ratio for the avoided toxicity 6 months after SBRT.
  The costs will be evaluated by the data from french social security system, from homogeneous group of patients and from general classification of professional acts
Cost/Efficacy ratio between 2 modalities of SBRT treatment of ependymoma at 12 months after treatment | 12 months after inclusion
  2 modalities of SBRT are compared in patients with an ependymoma (3 fractions of 8 Gy versus 5 fractions of 5 Gy). It will be calculated :
  * the cost/efficacity per gained year of life without relapse after 12 months after SBRT
  * the cost/efficacity per gained year of life without disease after 12 months after SBRT.
  The costs will be evaluated by the data from french social security system, from homogeneous group of patients and from general classification of professional acts
Cost/Efficacy ratio between 2 modalities of SBRT treatment of ependymoma at 24 months after treatment | 24 months after inclusion
  2 modalities of SBRT are compared in patients with an ependymoma (3 fractions of 8 Gy versus 5 fractions of 5 Gy). It will be calculated :
  * the cost/efficacity per gained year of life without relapse after 24 months after SBRT
  * the cost/efficacity per gained year of life without disease after 24 months after SBRT.
  The costs will be evaluated by the data from french social security system, from homogeneous group of patients and from general classification of professional acts

CONTACTS AND LOCATIONS:
Overall Officials: Line CLAUDE, Doctor, Principal Investigator — Centre Leon Berard
Locations (15):
- France (15):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - Centre Paul Strauss, Strasbourg, Bas-Rhin
  - Hôpital La Timone, Marseille, Bouches Du Rhône
  - Centre François Baclesse, Caen, Calvados
  - CHU Bordeaux - Hôpital Saint André, Bordeaux, Gironde
  - Centre Claudius Régaud, Toulouse, Haute Garonne
  - Institut de Cancérologie de Montpellier, Montpellier, Hérault
  - Centre Eugène Marquis, Rennes, Ille Et Vilaine
  - CHRU de Tours - Hôpital Bretonneau, Tours, Indre Et Loire
  - Institut de Cancérologie de l'Ouest René Gauducheau, Saint-Herblain, Loire Atlantique
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Centre Oscar Lambret, Lille, Nord
  - Centre Léon Bérard, Lyon, Rhône
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Institut Curie, Paris, Île-de-France Region

REFERENCES:
- [Background] Timmerman RD. An overview of hypofractionation and introduction to this issue of seminars in radiation oncology. Semin Radiat Oncol. 2008 Oct;18(4):215-22. doi: 10.1016/j.semradonc.2008.04.001. No abstract available. PMID 18725106
- [Background] Rapport ANAES : Evaluation clinique et économique de la radiochirurgie intra cranienne en conditions stéréotaxique - Rapport ANAES/Service évaluation des technologies-évaluation économique: 2000.
- [Background] Rapport HAS : Radiothérapie extra crânienne en conditions stéréotaxiques - Décembre 2006: 2006.
- [Background] Maranzano E, Anselmo P, Casale M, Trippa F, Carletti S, Principi M, Loreti F, Italiani M, Caserta C, Giorgi C. Treatment of recurrent glioblastoma with stereotactic radiotherapy: long-term results of a mono-institutional trial. Tumori. 2011 Jan-Feb;97(1):56-61. doi: 10.1177/030089161109700111. PMID 21528665
- [Background] Minniti G, Armosini V, Salvati M, Lanzetta G, Caporello P, Mei M, Osti MF, Maurizi RE. Fractionated stereotactic reirradiation and concurrent temozolomide in patients with recurrent glioblastoma. J Neurooncol. 2011 Jul;103(3):683-91. doi: 10.1007/s11060-010-0446-8. Epub 2010 Nov 5. PMID 21052773
- [Background] Torok JA, Wegner RE, Mintz AH, Heron DE, Burton SA. Re-irradiation with radiosurgery for recurrent glioblastoma multiforme. Technol Cancer Res Treat. 2011 Jun;10(3):253-8. doi: 10.7785/tcrt.2012.500200. PMID 21517131
- [Background] Zacharoulis S, Ashley S, Moreno L, Gentet JC, Massimino M, Frappaz D. Treatment and outcome of children with relapsed ependymoma: a multi-institutional retrospective analysis. Childs Nerv Syst. 2010 Jul;26(7):905-11. doi: 10.1007/s00381-009-1067-4. Epub 2009 Dec 29. PMID 20039045
- [Background] Kano H, Yang HC, Kondziolka D, Niranjan A, Arai Y, Flickinger JC, Lunsford LD. Stereotactic radiosurgery for pediatric recurrent intracranial ependymomas. J Neurosurg Pediatr. 2010 Nov;6(5):417-23. doi: 10.3171/2010.8.PEDS10252. PMID 21039163
- [Background] Liu AK, Foreman NK, Gaspar LE, Trinidad E, Handler MH. Maximally safe resection followed by hypofractionated re-irradiation for locally recurrent ependymoma in children. Pediatr Blood Cancer. 2009 Jul;52(7):804-7. doi: 10.1002/pbc.21982. PMID 19260098
- [Background] Combs SE, Behnisch W, Kulozik AE, Huber PE, Debus J, Schulz-Ertner D. Intensity Modulated Radiotherapy (IMRT) and Fractionated Stereotactic Radiotherapy (FSRT) for children with head-and-neck-rhabdomyosarcoma. BMC Cancer. 2007 Sep 13;7:177. doi: 10.1186/1471-2407-7-177. PMID 17854490
- [Background] Giller CA, Berger BD, Pistenmaa DA, Sklar F, Weprin B, Shapiro K, Winick N, Mulne AF, Delp JL, Gilio JP, Gall KP, Dicke KA, Swift D, Sacco D, Harris-Henderson K, Bowers D. Robotically guided radiosurgery for children. Pediatr Blood Cancer. 2005 Sep;45(3):304-10. doi: 10.1002/pbc.20267. PMID 15558704
- [Background] Grabb PA, Lunsford LD, Albright AL, Kondziolka D, Flickinger JC. Stereotactic radiosurgery for glial neoplasms of childhood. Neurosurgery. 1996 Apr;38(4):696-701; discussion 701-2. PMID 8692387
- [Background] Hodgson DC, Goumnerova LC, Loeffler JS, Dutton S, Black PM, Alexander E 3rd, Xu R, Kooy H, Silver B, Tarbell NJ. Radiosurgery in the management of pediatric brain tumors. Int J Radiat Oncol Biol Phys. 2001 Jul 15;50(4):929-35. doi: 10.1016/s0360-3016(01)01518-8. PMID 11429220
- [Background] Chawla S, Schell MC, Milano MT. Stereotactic body radiation for the spine: a review. Am J Clin Oncol. 2013 Dec;36(6):630-6. doi: 10.1097/COC.0b013e31822dfd71. PMID 22134513
- [Background] Lo SS, Sahgal A, Wang JZ, Mayr NA, Sloan A, Mendel E, Chang EL. Stereotactic body radiation therapy for spinal metastases. Discov Med. 2010 Apr;9(47):289-96. PMID 20423672
- [Background] Siva S, MacManus M, Ball D. Stereotactic radiotherapy for pulmonary oligometastases: a systematic review. J Thorac Oncol. 2010 Jul;5(7):1091-9. doi: 10.1097/JTO.0b013e3181de7143. PMID 20479693
- [Background] Fogh SE, Andrews DW, Glass J, Curran W, Glass C, Champ C, Evans JJ, Hyslop T, Pequignot E, Downes B, Comber E, Maltenfort M, Dicker AP, Werner-Wasik M. Hypofractionated stereotactic radiation therapy: an effective therapy for recurrent high-grade gliomas. J Clin Oncol. 2010 Jun 20;28(18):3048-53. doi: 10.1200/JCO.2009.25.6941. Epub 2010 May 17. PMID 20479391
- [Background] Flannery T, Kano H, Martin JJ, Niranjan A, Flickinger JC, Lunsford LD, Kondziolka D. Boost radiosurgery as a strategy after failure of initial management of pediatric primitive neuroectodermal tumors. J Neurosurg Pediatr. 2009 Mar;3(3):205-10. doi: 10.3171/2008.11.PEDS08268. PMID 19338466
- [Background] Conter C, Carrie C, Bernier V, Geoffray A, Pagnier A, Gentet JC, Lellouch-Tubiana A, Chabaud S, Frappaz D. Intracranial ependymomas in children: society of pediatric oncology experience with postoperative hyperfractionated local radiotherapy. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1536-42. doi: 10.1016/j.ijrobp.2008.09.051. Epub 2009 Apr 11. PMID 19362789
- [Background] Massimino M, Gandola L, Giangaspero F, Sandri A, Valagussa P, Perilongo G, Garre ML, Ricardi U, Forni M, Genitori L, Scarzello G, Spreafico F, Barra S, Mascarin M, Pollo B, Gardiman M, Cama A, Navarria P, Brisigotti M, Collini P, Balter R, Fidani P, Stefanelli M, Burnelli R, Potepan P, Podda M, Sotti G, Madon E; AIEOP Pediatric Neuro-Oncology Group. Hyperfractionated radiotherapy and chemotherapy for childhood ependymoma: final results of the first prospective AIEOP (Associazione Italiana di Ematologia-Oncologia Pediatrica) study. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1336-45. doi: 10.1016/j.ijrobp.2003.08.030. PMID 15050308
- [Background] Sharma MS, Kondziolka D, Khan A, Kano H, Niranjan A, Flickinger JC, Lunsford LD. Radiation tolerance limits of the brainstem. Neurosurgery. 2008 Oct;63(4):728-32; discussion 732-3. doi: 10.1227/01.NEU.0000325726.72815.22. PMID 18981883
- [Background] Merchant TE, Boop FA, Kun LE, Sanford RA. A retrospective study of surgery and reirradiation for recurrent ependymoma. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):87-97. doi: 10.1016/j.ijrobp.2007.09.037. PMID 18406885